CLINICAL TRIAL: NCT04720768
Title: A Phase 1B Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Combination of Encorafenib, Binimetinib and Palbociclib in Patients With BRAF-mutant Metastatic Melanoma (The CELEBRATE Study)
Brief Title: Encorafenib, Binimetinib and Palbociclib in BRAF-mutant Metastatic Melanoma CELEBRATE
Acronym: CELEBRATE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17/021
Record Dates: First submitted 2020-09-15; First posted 2021-01-22 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Metastasis
Keywords: BRAF-mutant positive
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — binimetinib; encorafenib; palbociclib

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase IB, non-randomised study consisting of a dose escalation phase and expansion phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose escalation phase (Experimental): Encorafenib (tablet) 450mg PO daily
  Binimetinib (tablet) 45mg PO BD
  Palbociclib (tablet) variable dose PO daily for 21 consecutive days on treatment, followed by 7 consecutive days off treatment in a 28 day cycle
  Interventions: Drug: Binimetinib; Drug: Encorafenib; Drug: Palbociclib

INTERVENTIONS:
Drug: Binimetinib — MEK inhibitor
Drug: Encorafenib — BRAF inhibitor
Drug: Palbociclib — CDK4/6 inhibitor

SUMMARY:
This is an open-label, phase IB, non-randomised study consisting of a dose escalation phase and expansion phase, evaluating the safety, tolerability and preliminary efficacy of the combination of encorafenib, binimetinib and palbociclib in patients with BRAF-mutant metastatic melanoma.

Dose escalation phase: Previously treated or treatment-naïve patients will be evaluated after the first cycle for dose-limiting toxicities to ascertain the recommended phase 2 dose (RP2D) of encorafenib, binimetinib and palbociclib.

Expansion phase: Two cohorts of patients will be further evaluated for the efficacy and safety of the RP2D of palbociclib with encorafenib and binimetinib. Cohort 1 will include patients naïve to both BRAF and MEK inhibitors. Cohort 2 will include patients with either primary or acquired resistance to both BRAF and MEK inhibitors.

DETAILED DESCRIPTION:
This is an open-label, multicentre, Phase IB, dose escalation study with dose expansion designed to assess the safety, tolerability, and pharmacokinetics of the encorafenib, binimetinib and palbociclib combination. Patients with untreated or previously treated BRAFV600 mutation-positive, locally advanced/unresectable or metastatic melanoma are eligible. There will be 3 dose levels:

Table 1: Dose Level Description Dose Level Encorafenib Binimetinib Palbociclib D1 450mg daily 45mg BID 75mg daily 21/7* D2 450mg daily 45mg BID 100mg daily 21/7* D3 450mg daily 45mg BID 125mg daily 21/7*

* 21 consecutive days on treatment, followed by 7 consecutive days off treatment in a 28 day cycle.

Alternate dosing regimens and schedules may be interrogated depending on the nature and timing of the toxicities encountered.

The first dose to be evaluated will be dose level D1 and dose escalation will follow using a standard 3 + 3 design (refer to Figure 6). Dose escalation/de-escalation decisions will be made by the Trial Management Committee.

Dose Limiting Toxicities (DLTs) will be monitored over the first 28 days of treatment. After each dose level of 3 patients complete the DLT observation period, the TMC will meet and review the available toxicity and dosing information and determine the dose regimen for the next dose level of 3 patients and/or identify the RP2D for the dose-expansion phase.

Approximately 30 additional patients will be enrolled into each of the two cohorts during the dose-expansion phase. One cohort will consist of previously untreated patients or treated patients without prior exposure to any BRAF and MEK inhibitor therapy. The second cohort will consist of patients who have progressed on BRAF and MEK inhibitor therapy.

A minimum of 10 patients in each cohort must have newly obtained tumour sample at baseline. Accrual may be restricted to achieve this. Treatment of patients in both phases will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion is met.

For the purpose of the final analyses, the study will be considered completed when 12 months have passed since the first day of treatment of the last patient enrolled in the expansion phase.

Adult patients with a diagnosis of BRAFV600 mutation positive, locally advanced/unresectable or metastatic melanoma who meet all the inclusion and none of the exclusion criteria will be eligible for participation in this study.

Recruitment will occur from all activated sites into the currently open phase and dose level of the study. Dose Level 1 will be the first to open and will enroll 3 patients at a minimum. The TMC will assess and determine the dose level for the next patients to open to recruitment accordly. Participants in the dose escalation phase will be evaluable for assessment if they complete 80% of their first cycle of combined treatment or they experience a DLT.

Once the RP2D has been determined by the TMC, recruitment will continue to occur from all activated sites into the dose expansion phase of the study. All patients in this phase will receive the RP2D. Patients in the dose expansion phase will be assigned to one of the 2 cohorts according to their treatment status (either BRAF/MEK-inhibitor naïve, or previously treated).

A number of assessments will occur while the patient is on treatment as well as the following:

PK sampling will be collected as part of the safety assessments according to the Schedule of Events in Section 3. On PK sampling days for trough levels (cycle 1 day 15 and cycle 2 day 1), study visits should be scheduled in the morning so a pre-dose PK blood sample can be collected. On these visit days, the morning dose of encorafenib, binimetinib and palbociclib will only be administered by the investigator (or designee) at the study site, after collecting the pre-dose PK sample. For PK visits, patients will be required to be fasting 2 hours before and 1 hour after the dose. Exact dates of drug administration (and actual PK blood draw) will be recorded on the appropriate eCRF. Any sampling problems (e.g. patient took study drug before draw took place) must be noted in the eCRF and on appropriate source documentation.

Tumour and blood samples collected for PD and biomarker assessments will be analysed with the objectives of understanding mechanisms of action and PD of the encorafenib, binimetinib and palbociclib combination, identifying biomarkers that are predictive of response, and explaining mechanisms of innate/acquired resistance.

Specimens for dynamic (non-inherited) and genetic (inherited) biomarkers will be collected from all patients on the trial.

Mandatory plasma samples will be collected from all patients, as described in the Schedule of Events. Circulating tumour DNA will be extracted and analysed for BRAF V600E and V600K mutation status. The mutation profile obtained from the circulating DNA will be compared with the mutation profile obtained from the tumour biopsy collected at baseline, during treatment and on progression. Plasma-circulating DNA carrying BRAF V600E mutation (BRAF-mutated alleles) will be detected and measured over time by determining percentages of total DNA and BRAF V600E concentration, either as relative percentage or absolute values. This may be useful to predict either disease progression at an early stage or response to therapy. The plasma samples may also be used to identify other potential predictive markers of clinical response to the encorafenib, binimetinib and palbociclib combination.

Whole blood sample will be analysed for mutations detected in tumour tissue, in order to verify the somatic nature of the mutations.

All patients will be required to provide newly collected tumour biopsies at baseline (unless inaccessible), on day 15 of cycle 1 and at the time of disease progression.

At least 2 cores per collection time point should be obtained (minimum of 1 core for FFPE, and if feasible, 1 core for fresh frozen biopsy). Excisional biopsies, punch biopsies and 14-gauge core needle biopsies are all acceptable. Fine needle aspiration biopsies will not be accepted.

Lesions with the greatest change in dimensional size, based on interval evaluation, are the lesions to be biopsied, if possible.

Scheduling of the on-treatment tumour biopsies should not interfere with the scheduling of the first, post-baseline FDG-PET scan. Ideally, tumour biopsies at screening and during Cycle 1 day 15 should be performed after the mandated FDG-PET scan.

The biopsy at disease progression should be taken from an enlarging lesion. Biopsies at progression should be obtained within 3 days of study drug discontinuation (i.e. continue study treatment for several days beyond documentation of progression, if necessary, in order to coordinate the timing of biopsy to occur within 3 days of study drug discontinuation).

FFPE tumour from baseline, on-treatment (Cycle 1 Day 15) and disease progression biopsies will be used to perform the following biomarker analyses:

* Immunohistochemistry (IHC) for molecules known to be relevant for activity of the MAPK and CDK4 pathways (e.g. ERK and MEK protein phosphorylation, RB1 phosphorylation).
* IHC for molecules that are potential PD biomarkers for encorafenib, binimetinib and palbociclib.
* IHC for molecules potentially related to response/resistance.
* Evaluation of the tumour microenvironment by multiplexed IHC and Nanostring gene-array technology.
* BRAF mutations (including V600E) and other somatic mutations.

Fresh-frozen tumour (baseline, Cycle 1 day 15, and at disease progression) may be used for whole genome analysis; other techniques such as reverse phase protein array or mRNA quantitation may also be performed.

There is increasing evidence that the gut microbiome plays a role in melanoma treatment outcome through its immune-modulating effects.

In this study, microbiome samples will be collected at baseline and at the end of treatment. DNA will be extracted from faecal samples. Gene sequencing will be performed to survey microbial species in the gut in order to define microbiota as a function of efficacy and safety. Overall changes in the gut microbiota will also be characterised in individual participants that receive therapy.

During the study, in addition to the biomarkers specified above, exploratory biomarker research may be conducted on any tumour (newly obtained or archival) and/or blood and/or plasma samples. These studies would extend the search for other potential biomarkers relevant to the effects of the drugs given in combination in this study, and/or prediction of these effects, and/or resistance to the treatment, and/or safety. This may also include research to help develop ways to detect, monitor or treat cancer. These additional investigations would be dependent upon clinical outcome, reagent and sample availability.

Patients enrolled in all phases of this study will be treated with the encorafenib, binimetinib and palbociclib combination until progression and/or experiencing unacceptable toxicity, and/or the treatment is discontinued at the discretion of the investigator or withdrawal of consent.

Treatment beyond progression of disease will be allowed only under special circumstances; for example: cystic lesions, mixed responses, and new brain metastasis which are treatable with stereotactic radiotherapy or surgery, but not requiring whole brain radiotherapy. It is judged by the investigator, in agreement with the CPI, whether or not a patient may remain on study treatment as long as he/she continues to benefit from the study drug treatment per investigator assessment. A treatment beyond progression consent form will not be required.

Tumour response will be evaluated locally by the investigator according to the RECIST version 1.1.

Patients will be evaluated for all potential sites of tumour lesions at Screening/baseline and every 8 weeks after starting study treatment until disease progression.

On-study tumour assessments have a ± 3-day window. There will be a tumour assessment at the 30 day safety follow-up (± 7 days) if the patient discontinues for any reason other than disease progression and the last tumour assessment has been performed > 28 days prior to this day.

Patients who discontinue study treatment due to a reason other than disease progression should continue to be followed and undergo tumour assessments every 8 weeks (± 3 days) until disease progression or initiation of subsequent anti-neoplastic therapy, or death, whichever occurs first.

Every effort must be made to assess each lesion that is measured at Screening/baseline by the same method throughout the study so that the comparison is consistent.

At all post-Screening/baseline assessments and the 30 day safety follow-up, the following should be performed:

* All patients are required to undergo chest, abdomen and pelvis CT/MRI scans.
* Brain MRI or CT scan, if metastases were documented at baseline
* Additional imaging evaluations may be performed at any time if there is symptomatic evidence suggesting the possibility of disease progression based on clinical symptoms or physical exam.

Criteria required for determining partial or complete response should be present for at least 4 weeks. All complete and partial responses must be confirmed by a second assessment at least 4 weeks later. If unscheduled imaging evaluations are performed (e.g. to confirm response or if progression is suspected), every effort should be made to perform subsequent imaging evaluations in accordance with the original imaging schedule. If evidence of progressive disease is nonequivocal, every effort should be made to keep the patient on study medication for at least one additional imaging evaluation as long as it is clinically acceptable.

CT scans should be acquired with IV contrast. If a patient is known to have a medical contraindication to CT IV contrast agent or develops a contraindication during the study, a CT scan without IV contrast of the chest and MRI with IV contrast, if possible, of the abdomen and pelvis may be performed. A CT scan of the brain, preferably with IV contrast, may be performed if MRI is contra-indicated.

Chest x-ray or ultrasound should not be used for tumour response assessments in this study.

Any lesions that have been subjected to loco-regional therapies (e.g., radiotherapy, ablation, etc.) should not be considered measurable, unless they have clearly progressed since the therapy. Previously treated lesions that have not progressed should be considered non-measurable and therefore, assessed as non-target lesions.

PET scan is not adequate for RECIST v1.1 response assessment. If a PET scan is used for determination of disease progression, then a corresponding CT and/or MRI scan is required. CT and/or MRI scans will be compared against PET scans.

Each centre should have a designated radiologist responsible for the interpretation of CT/MRI scans and response evaluations for study patients. Preferably, a single radiologist should perform all evaluations for an individual patient.

In this study, FDG-PET scans will be used to provide a non-invasive measurement of drug activity and a potential early readout of anti-tumour activity in patients on day 15 of Cycle 1. FDG-PET scans are optional for non-Australian sites. Metabolic response in a lesion will be assessed according to the method given in Wahl et al 2009 and will be centrally assessed at the Peter MacCallum Cancer Centre. Scans are read visually displayed side by side with liver uptake normalised between images. Response categories are defined as follows (comparison is with baseline PET scans in each case:

* Complete metabolic response (CMR): complete resolution of 18F-FDG uptake within measurable target lesion so that it is less than mean liver activity and indistinguishable from surrounding background blood-pool levels.
* Partial metabolic response (PMR): reduction of minimum of 30% in target measurable tumor 18F-FDG SUL peak. Absolute drop in SUL must be at least 0.8 SUL units, as well
* Stable metabolic disease (SMD): not CMR, PMR, or PMD.
* Progressive metabolic disease (PMD): 30% increase in 18F-FDG SUL peak, with .0.8 SUL unit increase in tumor SUV peak from baseline scan in pattern typical of tumor and not of infection/treatment effect. OR: Visible increase in extent of 18F-FDG tumor uptake (75% in TLG volume with no decline in SUL. OR: New 18F-FDG-avid lesions that are typical of cancer and not related to treatment effect or infection.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Phase only: (Australia only)

1. Patients who are naïve to, or have received prior BRAF and MEK inhibitor combination therapy. Prior treatment with chemotherapy and biological therapy (e.g. checkpoint inhibitor therapy) is permitted.

   Dose Expansion Phase only: (All sites)
2. Cohort 1: Patients who are naïve to BRAF and MEK inhibitor therapy. Prior treatment with chemotherapy and biological therapy (e.g. checkpoint inhibitor therapy) is permitted.
3. Cohort 2: Patients who have progressed on prior BRAF and MEK inhibitor combination therapy. Prior treatment with chemotherapy and biological therapy (e.g. checkpoint inhibitor therapy) is permitted.

   For both phases (All sites):
4. Patients (male and female) age ≥ 18 years
5. Has provided written informed consent prior to any screening procedure
6. Histologically confirmed diagnosis of unresectable stage III or IV melanoma (stage IIIB to IV per American Joint Committee on Cancer [AJCC] 8th edition).
7. Documented evidence of BRAF V600 mutation.
8. Patients must provide either archival or newly obtained tumour sample at baseline. In addition, patients must agree to a mandatory biopsy during treatment and at the time of progression, if not medically contraindicated.
9. Evidence of measurable disease, as determined by RECIST v1.1. Note: Lesions in areas of prior radiotherapy or other locoregional therapies (e.g., percutaneous ablation) should not be considered measurable, unless lesion progression has been documented since the therapy.
10. Patients must have adequate haematological, coagulation, renal and hepatic functions as defined by:

    Absolute neutrophil count ≥ 1.5 x 109/L Haemoglobin ≥ 10 g/L without transfusions Platelet count ≥ 100 x 109/L without transfusions Total serum creatinine ≤ 1.5 x ULN or calculated or directly measured CrCl < 50% LLN (lower limit of normal) Serum total bilirubin ≤ 1.5 x ULN ( 3 x ULN in cases of known Gilbert's syndrome) AST/SGOT or ALT/SGPT ˂ 3 x ULN, or ˂ 5 x ULN if liver metastases are present PT/INR or aPTT < 1.5xULN
11. ECOG Performance Status ≤ 2
12. Able to take oral medications
13. Be willing and able to comply with all study requirements, including treatment, attending assessments and follow-up.
14. Female patients of childbearing potential must have a negative serum pregnancy test at screening: and be willing to use two methods of birth control or be surgically sterile: or abstain from heterosexual activity for the course of the study through to 3 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilised or have not been free from menses for > 1 year.
15. Sexually active males must use a condom during intercourse while taking the study drugs and for 3 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomised men in order to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

1. Patients with uveal melanoma.
2. Patients with symptomatic or untreated brain metastases or leptomeningeal disease. Patients with previously treated or untreated for brain metastasis that are asymptomatic in the absence of corticosteroid therapy or on a stable dose of steroids for 4 weeks prior to registration are allowed to enroll. Brain metastases must be stable at least 4 weeks prior to registration with verification by imaging (e.g. brain MRI completed at screening demonstrating no current evidence of progressive brain metastases).
3. Patients receiving enzyme inducing anti-epileptic drugs (as listed in Appendix 5).
4. History of acute or chronic pancreatitis.
5. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
6. Impaired cardiovascular function or clinically significant cardiac disease including any of the following:

   * CHF requiring treatment (NYHA grade ≥ 2)
   * LVEF < 50% as determined by MUGA scan or ECHO
   * History or presence of clinically significant ventricular arrhythmias or uncontrolled atrial fibrillation
   * Clinically significant resting bradycardia
   * Unstable angina pectoris ≤ 3 months prior to registration
   * Acute Myocardial Infarction (AMI) ≤ 3 months prior to registration
   * QTcF > 480 ms
   * Any heart disease that requires the use of a cardiac pacemaker or implantable cardioverter defibrillator ≤ 3 months prior to registration
   * History of QT syndrome, Brugada syndrome or known

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLTs) | The assessment period of DLT for each patient is the first cycle (28 days) of treatment
  Dose-Limiting Toxicity is defined as a toxicity that prevents further administration of the trial treatment at that dose level

SECONDARY OUTCOMES:
Adverse events (AEs) of Encorafenib, Binimetinib and Palbociclib | Trough study completion, up until 12 months after last patient commences treatment
  Adverse events including type, grade and relationship to study treatment according to CTCAE v5.0
Tolerability as defined 80% compliance with each of Encorafenib, Binimetinib and Palbociclib individually. | 28 days for encorafenib and binimetinib, 21 days for palbociclib
  Tolerability: defined as ability to complete (with 80% compliance) cycle 1 of combination therapy. Compliance is defined as the percentage of days of treatment given at the assigned dose relative to the total number of days that treatment was intended to be given at the assigned dose (i.e. 28 days for encorafenib and binimetinib, 21 days for palbociclib). Eighty percent compliance must be achieved for each of the drugs considered separately for tolerability to be achieved.
Clinical effficacy defined by response | 8 weeks after commencement of treatment
  Clinical efficacy as defined by:
  o Best response at 8 weeks from start of treatment using RECIST v1.1 criteria
Clinical efficacy as defined by time to progression | From the date of registration until the date of disease progression
  Clinical efficacy as defined by:
  - Time to progression measured from the date of registration until the date of disease progression. Death, loss to follow up and follow up to the close out date without disease progression will be censoring events.
Clinical efficacy as defined by progression free survival | From the date of registration until the date of first documented disease progression or date of death due to any cause, whichever occurs first (up to approximately 18 months)
  Clinical efficacy as defined by:
  - Progression-free survival measured from the date of registration until the date of disease progression or the date of death from any cause. . Loss to follow up and follow up to the close out date without progression or death will be censoring events.
Clinical efficacy as defined by overall survival | From start of treatment until the date of death from any cause, up to approximately 18months)
  Clinical efficacy as defined by:
  - Overall survival measured from the date of registration until the date of death from any cause. Loss to follow up and follow up to the close out date without death will be censoring events.

OTHER OUTCOMES:
Response rates on Cycle 1 Day 15 | 8 weeks after commencement of treatment
  FDG-PET response rates on Cycle 1 Day 15
Mutation status of circulating DNA | From the date of registration to disease progression, up to approximately 18 months
  Mutational status of circulating tumour DNA at baseline, during treatment and at progression. Circulating tumour DNA will extracted and anakysed for BRAF V600E and V600K mutation status.
Genomic alterations in tumour tissue | From the date of registration to disease progression, up to approximately 18 months
  Genomic alterations in tumour tissue at baseline, on treatment and progression.Biomaker analyses to be performed include immunochemistry for molecules known to be relevant of the MAPK and CDK4 pathways, for molecules that are potential PD biomarkers for the trail drugs, potentially related to response/resistance, evaluation of the tumour microenvironment and BRAF mutations and other somatic mutations
Presence of biomarkers | From the time of screening, during treatment and 30 days after treatment
  Biomarkers in tumour tissue, blood and faecal microbiome for response/resistance

CONTACTS AND LOCATIONS:
Overall Officials: Grant McArthur, Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (4):
- Australia (4):
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data may be shared with external collaborators at other institutions. Any future data sharing agreement for future research will ensure data security and patient confidentiality in maintained.

REFERENCES:
- [Background] Ascierto PA, Dummer R, Gogas HJ, Flaherty KT, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, de Groot JWB, Loquai C, Gollerkeri A, Pickard MD, Robert C. Update on tolerability and overall survival in COLUMBUS: landmark analysis of a randomised phase 3 trial of encorafenib plus binimetinib vs vemurafenib or encorafenib in patients with BRAF V600-mutant melanoma. Eur J Cancer. 2020 Feb;126:33-44. doi: 10.1016/j.ejca.2019.11.016. Epub 2020 Jan 2. PMID 31901705
- [Background] Ascierto PA, Bechter O, Wolter P. A phase Ib/II dose-escalation study evaluation triple combination therapy with a BRAF (encorafenib), MEK (binimetinib), and CDK4/6 (ribociclib) inhibitor in patients with BRAF V600-mutant solid tumours and melanoma. J Clin Oncol. 2017;35 (suppl; abst 9518)
- [Background] Flaherty KT, Lorusso PM, Demichele A, Abramson VG, Courtney R, Randolph SS, Shaik MN, Wilner KD, O'Dwyer PJ, Schwartz GK. Phase I, dose-escalation trial of the oral cyclin-dependent kinase 4/6 inhibitor PD 0332991, administered using a 21-day schedule in patients with advanced cancer. Clin Cancer Res. 2012 Jan 15;18(2):568-76. doi: 10.1158/1078-0432.CCR-11-0509. Epub 2011 Nov 16. PMID 22090362